CLINICAL TRIAL: NCT03160053
Title: Improving Keloids Using Targeted Ultraviolet-B Irradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055540
Record Dates: First submitted 2017-04-07; First posted 2017-05-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Intervention Model Description: Each participant served as his/hers own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Keloids that were randomized to the treatment group, were exposed to Narrowband-UVB (NB-UVB). Targeted UVB will be delivered to the keloid for up to 16 weeks using the Lumera UVB light phototherapy device (Daavlin, Bryan Ohio, USA).The affected skin will be irradiated using a hand-held fiber optic cable with an adjustable aperture.
  Interventions: Device: NB-UVB
- Control Group (No Intervention): Keloids that were randomized to a non treatment group, were not exposed to the NB-UVB light.

INTERVENTIONS:
Device: NB-UVB — NB-UVB has an emission spectrum in the ultraviolet B range of 290-320 nm. The system consists of a light source, a spot handpiece, and a light guide that connects the handpiece to the light source. The light source has a Start/Stop switch for light beam activation. Activation can also be controlled remotely with a foot switch. The light source has a timer and an output level control to adjust the intensity of the ultraviolet light. This will be calibrated using a manufacturer-provided UV meter prior to every treatment to ensure accurate doses of ultraviolet light.
  Other Names: Narrowband UVB
  Arms: Treatment Group

SUMMARY:
Treatment of keloids with targeted Ultraviolet-Beta (UVB) radiation will improve the clinical appearance and induration of lesions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years old or over
* Participants must have a diagnosis of keloid
* No treatment with topical or intralesional steroids for 1 month prior to study

Exclusion Criteria:

* Patients who are unable to provide informed consent
* A history of photosensitivity, lupus erythematosus, porphyria or current use of a known photosensitizing drug
* Unwillingness to stop with topical or intralesional steroids for 1 month prior to study
* A history of malignant melanoma
* A history of radiation therapy to area of interest
* Subjects who self-report that they are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Clinical Appearance As Assessed by the Patient and Observer Scar Assessment (POSAS) Scale | 16 weeks
  Investigators will evaluate the pre- and post-study clinical photographs of all participants. The grading investigator will grade the degree of improvement using the POSAS scale to measure the clinical appearance of the keloids